CLINICAL TRIAL: NCT05947448
Title: Efficacy and Safety of Mexartan Potassium Tablets (AZL-M) and Calcium Channel Blockers (CCB) in the Treatment of Adults With Essential Hypertension in Chinese Population: a National Multicenter, Prospective, Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasten Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Ph4-HST-EDA-C-NIS-22-01
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-07

CONDITIONS: Essential Hypertension
Keywords: essential hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- AZL-M single drug group: Azilsartan Medoxomil Potassium Tablet，80mg，tablet，QD，six months
  Interventions: Drug: Azilsartan Medoxomil Potassium Tablet
- CCB single drug group: Nifedipine Controller-release Tablets，clinical maximum tolerated dose，tablet，QD，six months；or Levoamlodipine Maleate Table，clinical maximum tolerated dose，tablet，QD，six months； Doctor choose a medication that is more suitable for patient treatment.
  Interventions: Drug: Nifedipine Sustained -release Tablets; Drug: Levoamlodipine Maleate Table
- AZL-M + CCB drug group（Combined medication）: Nifedipine Controller-release Tablets，clinical maximum tolerated dose，tablet，QD，six months；and Levoamlodipine Maleate Table，clinical maximum tolerated dose，tablet，QD，six months； When the patient's upper pressure exceeds 160 Millimetre of mercury, the doctor will choose combination medication .CCB drug will be chosen either Nifedipine Controller-release Tablets or Levoamlodipine Maleate Table.
  Interventions: Drug: Azilsartan Medoxomil Potassium Tablet; Drug: Nifedipine Sustained -release Tablets; Drug: Levoamlodipine Maleate Table

INTERVENTIONS:
Drug: Azilsartan Medoxomil Potassium Tablet — Azilsartan Medoxomil Potassium Tablet，80mg，qd，lasts six month
  Groups: AZL-M + CCB drug group（Combined medication）; AZL-M single drug group
Drug: Nifedipine Sustained -release Tablets — Nifedipine Sustained -release Tablets，qd，The maximum clinical dose，lasts six months；
  Groups: AZL-M + CCB drug group（Combined medication）; CCB single drug group
Drug: Levoamlodipine Maleate Table — Levoamlodipine Maleate Table，qd，The maximum clinical dose，lasts six months；
  Groups: AZL-M + CCB drug group（Combined medication）; CCB single drug group

SUMMARY:
This is a national multicenter, prospective, observational study. It is planned to enroll 1215 patients with newly diagnosed essential hypertension in 80 centers, and divide them into 3 groups according to different treatment plans given by doctors: AZL-M monotherapy group, CCB monotherapy group (amlodipine besylate tablets or nifedipine controlled-release tablets) and AZL-M+CCB (amlodipine besylate tablets or nifedipine controlled-release tablets) combined treatment group. Subjects were visited 4 times at baseline, 1 month, 3 months, and 6 months, and the following key indicators of subjects were measured according to the doctor's decision, and the measurement results were collected

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old (one year old);
2. Patients diagnosed with essential hypertension;
3. Did not receive any antihypertensive drug treatment for at least 3 months before enrollment;
4. Eligible to use 80 mg once-daily AZL-M at baseline or CCB (amlodipine besylate tablets or nifedipine controlled-release tablets) or CCB (besylate Amlodipine tablets or nifedipine controlled-release tablets) + AZL-M 80 mg once-daily combination therapy; Volunteer to participate in this study, understand and sign the written informed consent.

Exclusion Criteria:

1. Used antihypertensive drugs for indications other than hypertension within 3 months before enrollment;
2. Has a history of alcoholism, drug abuse or illegal drug use;
3. Pregnant, breastfeeding women, and those who plan to become pregnant in the near future;
4. Life expectancy is less than one year; Participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: town hospital
Sampling Method: Non-Probability Sample
Enrollment: 1215 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the patient's blood pressure reached the target rate | 6 months
  Ø Compliance rate of systolic blood pressure (SBP) in the clinic: the proportion of subjects whose blood pressure dropped to sitting systolic blood pressure (sitSBP) <140 mmHg or compared with the baseline value of sitSBP ≥ 20mmHg;
  Ø Compliance rate of diastolic blood pressure (DBP) in the clinic: the proportion of subjects whose blood pressure dropped to sitting diastolic blood pressure (sitDBP) <90 mmHg or compared with the baseline value of sitDBP decreased by ≥10mmHg;
  Ø Achievement rate of both SBP and DBP in the clinic: the proportion of subjects who meet the SBP and DBP standards in the above clinics at the same time.

CONTACTS AND LOCATIONS:
Locations (1):
- Junbo Ge, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided